CLINICAL TRIAL: NCT01113970
Title: Phase I/II Study of a Novel Indibulin Dosing Schedule for the Treatment of Metastatic Breast Cancer
Brief Title: Study of a Novel Indibulin Dosing Schedule for the Treatment of Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL2001
Record Dates: First submitted 2010-04-08; First posted 2010-04-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; Indibulin; unresectable, locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — indibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): open label, single arm, unblinded
  Interventions: Drug: Indibulin

INTERVENTIONS:
Drug: Indibulin — Indibulin given orally once a day for 5 days followed by a 9 day rest
  Other Names: ZIO-301; Zybulin(TM)

SUMMARY:
This study is a Phase I/II trial of a novel Indibulin dosing schedule for the treatment of metastatic breast cancer. Eligible patients will have measurable or non-measurable, metastatic or unresectable, locally advanced breast cancer and may have received any number of prior therapies for their disease.

It is expected that the Phase I portion will enroll up to 20 patients and the Phase II portion will enroll up to 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of invasive carcinoma of the breast.
* Clinical evidence of metastatic disease or locally advanced disease not amenable to curative therapy.
* Measurable or non-measurable lesions according to the RECIST Version 1.1 2009.
* Any number of prior endocrine, biologic or chemotherapy regimens is permitted. All previous chemotherapy and biologic therapy must have been discontinued at least 3 weeks prior to beginning study drug. Endocrine therapy may not be used concurrently with protocol treatment. All acute toxic effects (excluding alopecia or neuropathy) of any prior therapy must have resolved to NCI CTC (version 4.0) Grade ≤ 1 or to baseline
* Prior radiation therapy is permitted.
* ECOG performance status of 0, 1 or 2.
* Age ≥ 18 years
* Life expectancy ≥ 12 weeks
* Patients with HER2-positive (IHC 3+ or FISH-amplified) breast cancer must have received trastuzumab or have a contradiction to receiving HER2- targeted therapy (such as abnormal left ventricular ejection fraction)as determined by the treating physician.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

  * Creatinine ≤ 1.5x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5x ULN
  * ALT or AST ≤ 2.5x ULN
  * ANC ≥ 1.5 x10(9)/L
  * Platelets ≥ 100 x10(9)/L
  * Hemoglobin ≥ 9g/dL
* Subjects of childbearing potential must agree to use a barrier method of contraception throughout the study and for 3 months after study drug administration.

Exclusion Criteria:

* Pregnant or nursing women may not participate.
* Serious, uncontrolled, concurrent infection.
* Patients with symptomatic CNS metastases that remain untreated by radiation therapy are excluded from this trial. The presence of asymptomatic, previously irradiated, stable brain metastases for at least 3 months are not grounds for trial exclusion.
* Presence of uncontrolled gastrointestinal malabsorption syndrome.
* Any chemotherapy, radiotherapy or breast cancer directed biologic therapy during the study or within 3 weeks of study start. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry. No washout period is required for hormonal therapies.
* Concurrent radiation therapy is not permitted during treatment on protocol.
* History of an invasive second primary malignancy diagnosed within the previous 3 years, except for Stage I endometrial or cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
* Any medical, psychological or social condition that may interfere with the subject's ability to safely participate in the study.
* Unwillingness to give written informed consent or unwillingness to participate or inability to comply with the protocol for the duration of the study. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures are necessary for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Phase I- Maximum Tolerated Dose | Throughout Cycle 1 (28 days)
  The primary objective of the Phase I portion of the trial is to determine the maximum tolerated dose (MTD) of Indibulin when given for 5 days followed by a 9 day rest (5-9) using a standard 3+3 dose escalation scheme for the treatment of metastatic breast cancer
Phase II- Progression Free Survival | 4 months
  The primary objective of the Phase II portion of this trial is to examine the efficacy of indibulin for the treatment of metastatic breast cancer at the MTD established in Phase I. The primary endpoint is the proportion of patients who are progression free at 4 months when treated with Indibulin (5-9)at the MTD determined by the phase I portion of the trial.

SECONDARY OUTCOMES:
Phase I- Number of participants with Adverse Events as a measure of safety and tolerability | Duration of study, approximately one year
  To evaluate the safety of Indibulin when administered for 5 days followed by a 9 day rest (5-9) in patients with metastatic breast cancer
Phase I- Toxicity | Cycle 1 (28 days), and duration of study (approximately one year)
  To describe the Cycle I and overall toxicity rates of indibulin (5-9) using the NCI CTC version 3.
Phase I- Pharmacokinetics of indibulin in study subject plasma assessed in Cycle 1 Day 1 and Cycle 1 Day 5 per schedule below in Description section. | During Cycle 1 (28 days)
  To evaluate pharmacokinetics (PK) of Indibulin (5-9) as it is assessed in Cycle 1 Day 1, Day 2, Day 5 and Day 8. Cycle 1 PK schedule as follows: Day 1 immediately pre dose, 1 hour, 2 hours, 4 hours, 6 hours and approximately 24 hours after start of infusion (Cycle 2 Day 1), Day 5 pre-dose and at anytime during Day 8.
Phase II- Overall Response Rate | At the end of Cycles 4 and 6 (approximately 4 months and 6 months respectively)
  To estimate the overall response rate (complete response and partial response)associated with Indibulin (5-9) schedule at eth MTD determined by the Phase I portion of this trial in patients with metastatic breast cancer.
Phase II- Rate of Stable Disease | Phase II- greater than 6 months
  To estimate the rate of stable disease greater than 6 months associated with the Indibulin (5-9) schedule at the MTD determined by the the Phase I portion of this trial in patients with metastatic breast cancer.
Phase II- Number of patients with Adverse Events as a measure of safety and tolerability | Throughout study, approximately one year
  To evaluate the safety of Indibulin when administered for 5 days followed by a 9 day rest (5-9) at the MTD determined by the Phase I portion of this trial in patients with metastatic breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J. Lewis, MD, PhD, Study Director — ZIOPHARM, Oncology, Inc.
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The West Clinic, Memphis, Tennessee
  - Evergreen Hematology Oncology, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268
- See also: ZIOPHARM Oncology, Inc. home page — http://www.ziopharm.com